CLINICAL TRIAL: NCT02360670
Title: Penumbra and Recanalisation Acute Computed Tomography in Ischaemic Stroke Evaluation
Acronym: PRACTISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); University of Edinburgh (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GN11NE418
Record Dates: First submitted 2015-01-21; First posted 2015-02-10 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Ischaemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control imaging (NCCT) (Placebo Comparator): Standard imaging
  Interventions: Other: control imaging
- additional multimodal imaging (Experimental): CT + CTA + CTP
  Interventions: Other: additional multimodal imaging

INTERVENTIONS:
Other: control imaging
  Arms: Control imaging (NCCT)
Other: additional multimodal imaging
  Arms: additional multimodal imaging

SUMMARY:
Stroke affects over 125,000 people each year in the UK and leaves at least 50% disabled. Treatment of stroke caused by a blockage in a blood vessel (ischaemic stroke), with clotbusting drugs improves the chances of good recovery, but must be given within 4.5 hours of onset. Currently only a small proportion of patients who arrive in hospital within 4.5 hours are treated. This is largely due to uncertainty about diagnosis and concerns about risk of bleeding associated with clotbusting medication. Patients with mild or improving symptoms in particular are often not treated because of uncertainty about relative risks and benefits. However, around one third of these patients go on to be significantly disabled. Routine CT scanning often does not show abnormalities in acute stroke (which take hours to become easily visible), and cannot show the extent or severity of blood flow changes in ischemic stroke.

We wish to investigate the value of additional CT scanning that gives information on the blood vessels (angiography, CTA) and blood flow to the brain (perfusion, CTP) by undertaking a randomised trial. Extra scans are done in the same scanner and involve some extra radiation, injections of a contrast dye, and some extra time to acquire process and interpret. The extra scans may allow better treatment decisions for patients by increasing diagnostic certainty and by better assessment of stroke severity. However, we do not know whether the potential gains from better selection justify the resources and potential treatment delays that are involved. We will investigate whether the proportion of patients given clotbusting drugs differs between the two scanning protocols; and whether the outcomes differ, using standard measures of disability. We will also investigate whether use of different scanner manufacturers' software affect interpretation of scans.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke eligible for IV rtPA according to current guidelines
* Informed consent
* Male or nonpregnant female ≥18 years of age
* Within 4.5 hours of onset as defined by time since last known well

Exclusion Criteria:

* Contraindications to thrombolytic drug treatment for stroke
* Pregnancy
* Known impaired renal function precluding contrast CT
* Known allergy to CT contrast agents
* Severe concurrent medical condition that would prevent participation in study procedures (e.g. cardiac failure with severe pulmonary oedema) or with life expectancy ≤ 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-08-26 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving Intravenous Recombinant Tissue Plasminogen Activator (IV rtPA) | 4.5 hours from onset
  Data will be collected at 4.5 hours from onset, comparison of proportion of patients receiving treatment will only be assessed at the end of the study

SECONDARY OUTCOMES:
Time to treatment decision and administration | 4.5 hours from onset
3 month modified Rankin Scale (mRS), by intention to treat, using a Cochran Mantel Haeszel distribution analysis | 90 days from onset
Safety - symptomatic Intracerebral hemorrhage (ICH) and major infarct swelling rates | 7 days from onset
Diagnostic sensitivity and specificity | 4.5 hours from onset
  Data will be collected at 4.5 hours from onset, comparison of proportion of patients receiving treatment will only be assessed at the end of the study
3 month mRS distribution in patients i) selected for IV rtPA and excluded from IV rtPA | 90 days from onset
Comparisons of efficacy & safety outcomes in Target Population (imaged as per randomised allocation and per protocol) | 90 days after onset
  Data will for safety will be collected at day 7, data for efficacy will be collected at day 90. Comparison between to groups will be done at the end of the study
Interobserver Agreement for rtPA eligibility between local and centrally processed CTP/CTA | Six months after recruitment
  Scans will be collected, centrally processed and presented again to the local clinicians in electronic form. Participants will be asked about clinical decision in view of centrally processed scans. The final data about inter observer agreement will be available at the end of the study
Interobserver agreement in interpretation of locally processed Computed Tomography Perfusion (CTP) scans | Six months after recruitment
  Scans will be collected, centrally processed and presented again to the clinicians in electronic form. The final data about inter observer agreement will be available at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Keith Muir, MBChB, MSc, MD, FRCP, Principal Investigator — University of Glasgow
Locations (1):
- Southern General Hospital, NHS Greater Glasgow and Clyde, Glasgow, United Kingdom